CLINICAL TRIAL: NCT00416650
Title: Multicenter Phase II Trial of OSI-774 (Erlotinib, Tarceva) in Patients With Advanced Bronchioalveolar Cell Lung Cancer.
Brief Title: Erlotinib in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Pao, MD, Professor of Medicine, Cancer Biology, & Pathology/ Microbiology/ Immunology; Director, Division of Hematology and Oncology; Ingram Professor of Cancer Research; Director, Personalized Cancer Medicine; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCC THO 0214; P50CA090949 (NIH); P30CA068485 (NIH); VU-VCC-THO-0214; VU-VCC-IRB-02-0168; GENENTECH-VU-VCC-THO-0214
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; bronchoalveolar cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental): Patients will receive erlotinib (OSI-774) 150 mg daily by mouth. If specified toxicities occurs, the dose may be reduced.
  Interventions: Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — All patients will receive 150 mg orally daily
  Other Names: Tarceva, OSI-774

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the major objective response rate (partial response and complete response) in patients with advanced bronchoalveolar cell non-small cell lung cancer treated with erlotinib hydrochloride.

Secondary

* Assess the quality of life of patients treated with this regimen.
* Determine the duration of response and time to disease progression in patients treated with this regimen.
* Determine the median survival of patients treated with this regimen.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive oral erlotinib hydrochloride daily in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed bronchoalveolar cell (or a variant) non-small cell lung cancer (NSCLC)

  * Stage IIIB (malignant pleural or pericardial effusion) disease
  * Stage IV disease
  * Recurrent and/or medically inoperable disease
* Measurable or evaluable indicator lesions
* No uncontrolled CNS metastases (i.e., any known CNS lesion that is radiographically unstable, symptomatic, and/or requiring escalating doses of corticosteroids)

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 80-100%
* Life expectancy ≥ 8 weeks
* WBC ≥ 3,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.0 mg/dL
* AST ≤ 2 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 55 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No significant medical history or unstable medical condition, including any of the following:

  * Unstable systemic disease
  * Congestive heart failure
  * Recent myocardial infarction
  * Unstable angina
  * Active infection
  * Uncontrolled hypertension
* No other active malignancies within the past 5 years except for adequately treated carcinoma of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior radiation therapy to a major bone marrow-containing area
* At least 3 weeks since prior chemotherapy
* No more than 1 prior chemotherapy regimen for NSCLC
* No prior systemic cytotoxic chemotherapy for other malignant diseases
* No prior erlotinib hydrochloride or other agents targeting the HER family (e.g., cetuximab, trastuzumab [Herceptin®], or gefitinib)
* No concurrent radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-07; Primary Completion 2007-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Major objective response rate (complete response and partial response) | At 4 weeks and then every 8 weeks
  Per Response Evaluation in Solid Tumors (RECIST) criteria v. 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions

SECONDARY OUTCOMES:
Worst grade toxicity | weekly for 4 weeks, then every 8 weeks to discontinuation of drug
  Number of patients with worst-grade toxicity at each of five grades (1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, disabling, 5 = death) following NCI Common Toxicity Criteria, v. 2. Drug is discontinued for disease progression, unacceptable toxicity, patient undergoes radiation or other chemotherapy, or withdraws from study
Quality of life as measured by the Lung Cancer Symptom Scale for patients | baseline, every week for 5 weeks, and then every 4 weeks
  The Lung Cancer Symptom Scale for patients is a nine-item scale with 0 = lowest rating (least) to 100 = highest rating (worst) for the measurement of symptom burden for loss of appetite, fatigue, cough, dyspnea, hemoptysis, activity, quality of life, lung cancer symptoms, and pain.
Survival | from study entry to date of death or last date known alive
  Duration of time from date of study entry to death from any cause or to the last date the patient is known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: William Pao, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas